CLINICAL TRIAL: NCT01956500
Title: Influence of Instaflex Joint Support Supplement on Joint Pain, Stiffness, Function, and Inflammation: a Randomized, Placebo-controlled Community Trial
Brief Title: Instaflex and Joint Pain in Community Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Collaborators: Direct Digital (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-0173
Record Dates: First submitted 2013-09-27; First posted 2013-10-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Joint Pain, Stiffness, Function
Keywords: glucosamine; inflammation; quality of life; physical function
MeSH Terms: conditions — Arthralgia; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Instaflex (Experimental): Instaflex Joint Support supplement (3 capsules per day for 8 weeks)
  Interventions: Dietary Supplement: Instaflex
- Placebo (Placebo Comparator): Placebo (3 capsules per day for 8 weeks)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Instaflex — The Instaflex supplement contained the following ingredients (in 3 capsules): Glucosamine sulfate (1500 mg), methylsulfonylmethane (MSM) (500 mg), white willow bark extract (standardized to 15% salicin) (250 mg), ginger root concentrate (50 mg), boswella serrata extract (standardized to 65% boswellic acid) (125 mg), turmeric root extract (50 mg), cayenne 40m H.U. (50 mg), and hyaluronic acid (4.0 mg).
  Other Names: Instaflex Joint Support dietary supplement
  Arms: Instaflex
Dietary Supplement: Placebo — The placebo capsules will contain magnesium stearate, an inert substance.
  Other Names: Placebo supplement
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to assess the effect of 8-weeks ingestion of the Instaflex Joint Support supplement (Direct Digital, Charlotte, NC) compared to placebo on joint pain, stiffness, and function (questionnaires and 6-min walk test) and blood inflammation biomarkers in adults with self-reported joint pain.

DETAILED DESCRIPTION:
Allocation: Randomized. Subjects will be randomized to one of two groups: placebo or Instaflex Joint Support. Supplements will be administered in double-blinded fashion.

Intervention Model: Instaflex Joint Support supplement for 8 weeks versus placebo.

Sample Size: N=100, with N=50 per group.

Statistical Procedures: 2 x 2 repeated measures analysis of variance (ANOVA).

Study Duration (per subject): 8 weeks.

Blood sample schedule: Blood draws pre- and post-study.

Monitoring adverse events: Subjects will fill in bi-weekly symptom logs to monitor untoward symptoms. Diagnostic chemistry panels will be measured pre- and post-study.

Rescue medication: Paracetamol (i.e., acetaminophen as found in Tylenol) will be allowed as a rescue medicine for pain during the study as needed. Subjects will record paracetamol usage. Paracetamol can relieve pain in mild arthritis but has no effect on the underlying inflammation, redness, and swelling of the joint.

Lab visit testing sequence (at the Kannapolis YMCA, in the afternoon by appointment.):

1. First visit:

   1. Consent form
   2. Medical health questionnaire to verify medical history, and lifestyle habits.
   3. Symptoms log for previous 2-weeks symptomatology
   4. Height, weight, and percent body fat (bioelectrical impedance, Tanita scale)
   5. Questionnaires: Western Ontario and McMaster Universities Arthritis Index (WOMAC), Short Form (36) Health Survey (SF-36), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP).
   6. Blood sample (followed by a glass of orange juice)
   7. 6-minute walk test (at the local YMCA track) (one practice trial, and then repeat for test).
   8. Receive supplement organizer tray with 8-weeks supply (and instructions)
2. 8-week study:

   a. Subjects will be contacted via email every 2 weeks to monitor compliance and fill in symptom logs.
3. Second lab visit:

   1. Same as first lab visit, except for removal of steps "a,b, and h".

Supplements:

Supplements (Instaflex, placebo) will be prepared in colored gel capsules (3 per day, identical looking), and given to the subjects in supplement organizer trays. Subjects will take 3 capsules/day: one capsule each in the morning, at noontime, and in the evening. The placebo capsules will contain magnesium stearate, an inert substance.

Compliance:

Compliance will be monitored with bi-weekly email messages, and by counting unused capsules when subjects return the supplement trays at the end of the 8-week study. If subjects miss one, two, or three days of taking supplements, subjects will be asked to double up usage until back on schedule. Subjects missing more than three days of taking the supplements will be asked to leave the study.

1. Instaflex Joint Support Supplement

A serving size is 3 capsules, and contains the following ingredients:

Glucosamine Sulfate 1500 mg Methylsulfonylmethane 500 mg White Willow Bark Extract (standardized to 15% salicin) 250 mg Ginger Root Concentrate 50 mg Boswella Serrata Extract (Standardized to 65% boswellic acid) 125 mg Turmeric Root Extract 50 mg Cayenne 40m H.U. 50 mg Hyaluronic Acid 4.0 mg Other Ingredients: Rice Flour, Gelatin, Vegetable Magnesium Stearate, Silicon Dioxide

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* ages 50-75 years
* history (>3 months) joint pain, knees, hip, ankles, shoulders, or hands
* willingness to avoid NSAIDs use during the 8-week study
* willingness to avoid other anti-inflammatory medications
* agree to stay weight stable during the 8-week study
* willing to follow all study procedures, including randomization to one of two groups
* able to walk for at least 6 min at a moderate-to-brisk pace

Exclusion Criteria:

* history of regular NSAID use during the previous two weeks
* use of other medications (e.g., analgesic gels, arthritis medications, other anti-inflammatory drugs) or supplements (in particular, glucosamine and chondroitin) for joint pain for the previous two weeks
* serious medical problems (current cancer case, severe rheumatoid arthritis, recent heart attack, recent stroke, congestive heart failure, ulcers, kidney disease, or other disease that will interfere with study participation).
* psychiatric disorder or other condition that might interfere with self-assessment ability.
* history of allergic reactions to shellfish products.
* history of allergic reactions to products containing aspirin.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Joint pain and function | Change in joint pain and function at 8 weeks
  Assessed through questionnaires

SECONDARY OUTCOMES:
Systemic inflammation | Change in systemic inflammation at 8 weeks
  Serum CRP and plasma cytokines (9 total)
Safety | Change in safety outcomes at 8 weeks
  Symptoms logs and diagnostic chemistries

CONTACTS AND LOCATIONS:
Overall Officials: David C. Nieman, DrPH, Principal Investigator — Appalachian State University
Locations (1):
- ASU Human Performance Laboratory, North Carolina Research Campus, Kannapolis, North Carolina, United States

REFERENCES:
- [Derived] Nieman DC, Shanely RA, Luo B, Dew D, Meaney MP, Sha W. A commercialized dietary supplement alleviates joint pain in community adults: a double-blind, placebo-controlled community trial. Nutr J. 2013 Nov 25;12(1):154. doi: 10.1186/1475-2891-12-154. PMID 24274358
- See also: Lab web site — http://www.ncrc.appstate.edu